CLINICAL TRIAL: NCT01389843
Title: Registry (Prospective Cohort) for Heart Failure in Korea (KorAHF)
Acronym: KorAHF
Status: Completed | Type: Observational
Sponsor: Byung-Hee Oh (Other)
Collaborators: National Institute of Health, Korea (Other Government)
Responsible Party: Sponsor-Investigator, Byung-Hee Oh, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Other Study IDs: H-1102-072-352
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Heart failure; Registry; Cohort; Heart Disease; Cardiovascular Diseases
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All consecutive hospitalized adult patients: All consecutive hospitalized adult patients who have 1 and (2 and/or 3)
  1. Symptom and/or sign of heart failure
  2. Lung congestion
  3. Objective finding of LV systolic dysfunction (LVEF), or structural heart disease.

SUMMARY:
KorAHF is a multi-center registry (prospective cohort) for acute decompensated heart failure patients in Korea.

The aim of this registry is to analyze several causes affecting prognosis and survival and to develop new strategies for managing acute decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

All consecutive hospitalized adult patients who have 1 and (2 and/or 3)

1. Symptom and/or sign of heart failure
2. Lung congestion
3. Objective finding of LV systolic dysfunction (LVEF), or structural heart disease

Exclusion Criteria:

* N.C.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: acute decompensated heart failure
Sampling Method: Non-Probability Sample
Enrollment: 5625 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Mortality and Re-hospitalization of acute decompensated heart failure | 5 years (tentative)
  1. In-hospital mortality
  2. Annual mortality
  3. Re-hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Hee Oh, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Data be shared with participating institution and NNIH

REFERENCES:
- [Derived] Yoon M, Park JJ, Youn JC, Lee SE, Lee HY, Choi JO, Kim KH, Yang DH, Cho MC, Kang SM, Yoo BS. Comparison of Natriuretic Peptide Levels in Sinus Rhythm and Atrial Fibrillation in Acute Heart Failure. Int J Heart Fail. 2025 Apr 24;7(2):85-95. doi: 10.36628/ijhf.2025.0007. eCollection 2025 Apr. PMID 40519716
- [Derived] Cho Y, Yoon M, Kim J, Lee JH, Oh IY, Lee CJ, Kang SM, Choi DJ. Artificial Intelligence-Based Electrocardiographic Biomarker for Outcome Prediction in Patients With Acute Heart Failure: Prospective Cohort Study. J Med Internet Res. 2024 Jul 3;26:e52139. doi: 10.2196/52139. PMID 38959500
- [Derived] Kim ES, Park SK, Youn JC, Lee HS, Lee HY, Cho HJ, Choi JO, Jeon ES, Lee SE, Kim MS, Kim JJ, Hwang KK, Cho MC, Chae SC, Kang SM, Park JJ, Choi DJ, Yoo BS, Cho JY, Kim KH, Oh BH, Greenberg B, Baek SH. Real-World Eligibility and Cost-Effectiveness Analysis of Empagliflozin for Heart Failure in Korea. J Korean Med Sci. 2024 Jan 8;39(1):e8. doi: 10.3346/jkms.2024.39.e8. PMID 38193327
- [Derived] Hong JA, Kim MS, Park H, Lee SE, Lee HY, Cho HJ, Choi JO, Jeon ES, Hwang KK, Chae SC, Baek SH, Kang SM, Choi DJ, Yoo BS, Kim KH, Cho MC, Kim JJ, Oh BH. Prognostic Value of QRS Duration among Patients with Cardiogenic Shock Complicating Acute Heart Failure: Data from the Korean Acute Heart Failure (KorAHF) Registry. Int J Heart Fail. 2020 Mar 16;2(2):121-130. doi: 10.36628/ijhf.2019.0016. eCollection 2020 Apr. PMID 36263287
- [Derived] Park J, Mebazaa A, Park JJ, Rhee TM, Park HA, Lee GY, Choi JO, Jeon ES, Lee SE, Cho HJ, Lee HY, Oh BH, Choi DJ; Korean Acute Heart Failure (KorAHF) Investigators. Incidence, Risk Factors and Prognosis of Contrast-Induced Acute Kidney Injury in Acute Heart Failure Patients Undergoing Coronary Angiography. Int J Heart Fail. 2019 Oct 24;1(1):72-85. doi: 10.36628/ijhf.2019.0006. eCollection 2019 Oct. PMID 36262741
- [Derived] Kim W, Park JJ, Lee HY, Kim KH, Yoo BS, Kang SM, Baek SH, Jeon ES, Kim JJ, Cho MC, Chae SC, Oh BH, Kook W, Choi DJ. Predicting survival in heart failure: a risk score based on machine-learning and change point algorithm. Clin Res Cardiol. 2021 Aug;110(8):1321-1333. doi: 10.1007/s00392-021-01870-7. Epub 2021 Jul 14. PMID 34259921
- [Derived] Park JJ, Lee HY, Kim KH, Yoo BS, Kang SM, Baek SH, Jeon ES, Kim JJ, Cho MC, Chae SC, Oh BH, Choi DJ. Heart failure and atrial fibrillation: tachycardia-mediated acute decompensation. ESC Heart Fail. 2021 Aug;8(4):2816-2825. doi: 10.1002/ehf2.13354. Epub 2021 May 6. PMID 33960144
- [Derived] Cho Y, Cho SY, Oh IY, Lee JH, Park JJ, Lee HY, Kim KH, Yoo BS, Kang SM, Baek SH, Jeon ES, Kim JJ, Cho MC, Chae SC, Oh BH, Choi DJ. Implantable Cardioverter-defibrillator Utilization and Its Outcomes in Korea: Data from Korean Acute Heart Failure Registry. J Korean Med Sci. 2020 Nov 30;35(46):e397. doi: 10.3346/jkms.2020.35.e397. PMID 33258331
- [Derived] Park CS, Park JJ, Mebazaa A, Lee HY, Kim KH, Yoo BS, Kang SM, Baek SH, Jeon ES, Kim JJ, Cho MC, Chae SC, Oh BH, Choi DJ. Response to beta-blockers and natriuretic peptide level in acute heart failure: analysis of data from the Korean acute heart failure registry. Clin Res Cardiol. 2021 Sep;110(9):1392-1403. doi: 10.1007/s00392-020-01689-8. Epub 2020 Jun 25. PMID 32588127
- [Derived] Kong MG, Jang SY, Jang J, Cho HJ, Lee S, Lee SE, Kim KH, Yoo BS, Kang SM, Baek SH, Choi DJ, Jeon ES, Kim JJ, Cho MC, Chae SC, Oh BH, Lim S, Park SK, Lee HY. Impact of diabetes mellitus on mortality in patients with acute heart failure: a prospective cohort study. Cardiovasc Diabetol. 2020 May 2;19(1):49. doi: 10.1186/s12933-020-01026-3. PMID 32359358
- [Derived] Son MK, Park JJ, Lim NK, Kim WH, Choi DJ. Impact of atrial fibrillation in patients with heart failure and reduced, mid-range or preserved ejection fraction. Heart. 2020 Aug;106(15):1160-1168. doi: 10.1136/heartjnl-2019-316219. Epub 2020 Apr 27. PMID 32341140
- [Derived] Seo WW, Park JJ, Park HA, Cho HJ, Lee HY, Kim KH, Yoo BS, Kang SM, Baek SH, Jeon ES, Kim JJ, Cho MC, Chae SC, Oh BH, Choi DJ. Guideline-directed medical therapy in elderly patients with heart failure with reduced ejection fraction: a cohort study. BMJ Open. 2020 Feb 6;10(2):e030514. doi: 10.1136/bmjopen-2019-030514. PMID 32034017
- [Derived] Park JJ, Park CS, Mebazaa A, Oh IY, Park HA, Cho HJ, Lee HY, Kim KH, Yoo BS, Kang SM, Baek SH, Jeon ES, Kim JJ, Cho MC, Chae SC, Oh BH, Choi DJ. Characteristics and outcomes of HFpEF with declining ejection fraction. Clin Res Cardiol. 2020 Feb;109(2):225-234. doi: 10.1007/s00392-019-01505-y. Epub 2019 Jul 2. PMID 31267239
- [Derived] Lee JH, Park JJ, Cho Y, Oh IY, Yoo BS, Kim JJ, Kim KH, Kang SM, Baek SH, Jeon ES, Cho MC, Chae SC, Oh BH, Choi DJ. Prognostic Implication of Ventricular Conduction Disturbance Pattern in Hospitalized Patients with Acute Heart Failure Syndrome. Korean Circ J. 2019 Jul;49(7):602-611. doi: 10.4070/kcj.2018.0290. Epub 2019 Feb 26. PMID 30891964
- [Derived] Park CS, Park JJ, Mebazaa A, Oh IY, Park HA, Cho HJ, Lee HY, Kim KH, Yoo BS, Kang SM, Baek SH, Jeon ES, Kim JJ, Cho MC, Chae SC, Oh BH, Choi DJ. Characteristics, Outcomes, and Treatment of Heart Failure With Improved Ejection Fraction. J Am Heart Assoc. 2019 Mar 19;8(6):e011077. doi: 10.1161/JAHA.118.011077. PMID 30845873
- [Derived] Park JJ, Park HA, Cho HJ, Lee HY, Kim KH, Yoo BS, Kang SM, Baek SH, Jeon ES, Kim JJ, Cho MC, Chae SC, Oh BH, Choi DJ. beta-Blockers and 1-Year Postdischarge Mortality for Heart Failure and Reduced Ejection Fraction and Slow Discharge Heart Rate. J Am Heart Assoc. 2019 Feb 19;8(4):e011121. doi: 10.1161/JAHA.118.011121. PMID 30755071
- [Derived] Choi KH, Han S, Lee GY, Choi JO, Jeon ES, Lee HY, Lee SE, Kim JJ, Chae SC, Baek SH, Kang SM, Choi DJ, Yoo BS, Kim KH, Cho MC, Park HY, Oh BH. Prognostic Significance of Left Axis Deviation in Acute Heart Failure Patients with Left Bundle branch block: an Analysis from the Korean Acute Heart Failure (KorAHF) Registry. Korean Circ J. 2018 Nov;48(11):1002-1011. doi: 10.4070/kcj.2018.0048. PMID 30334387
- [Derived] Lee SE, Lee HY, Cho HJ, Choe WS, Kim H, Choi JO, Jeon ES, Kim MS, Hwang KK, Chae SC, Baek SH, Kang SM, Choi DJ, Yoo BS, Kim KH, Cho MC, Kim JJ, Oh BH. Coronary artery bypass graft versus percutaneous coronary intervention in acute heart failure. Heart. 2020 Jan;106(1):50-57. doi: 10.1136/heartjnl-2018-313242. Epub 2018 Sep 12. PMID 30209124
- [Derived] Park JJ, Kim SH, Oh IY, Choi DJ, Park HA, Cho HJ, Lee HY, Cho JY, Kim KH, Son JW, Yoo BS, Oh J, Kang SM, Baek SH, Lee GY, Choi JO, Jeon ES, Lee SE, Kim JJ, Lee JH, Cho MC, Jang SY, Chae SC, Oh BH. The Effect of Door-to-Diuretic Time on Clinical Outcomes in Patients With Acute Heart Failure. JACC Heart Fail. 2018 Apr;6(4):286-294. doi: 10.1016/j.jchf.2017.12.017. PMID 29598933
- [Derived] Kang J, Park JJ, Cho YJ, Oh IY, Park HA, Lee SE, Kim MS, Cho HJ, Lee HY, Choi JO, Hwang KK, Kim KH, Yoo BS, Kang SM, Baek SH, Jeon ES, Kim JJ, Cho MC, Chae SC, Oh BH, Choi DJ. Predictors and Prognostic Value of Worsening Renal Function During Admission in HFpEF Versus HFrEF: Data From the KorAHF (Korean Acute Heart Failure) Registry. J Am Heart Assoc. 2018 Mar 13;7(6):e007910. doi: 10.1161/JAHA.117.007910. PMID 29535141
- [Derived] Lee SE, Lee HY, Cho HJ, Choe WS, Kim H, Choi JO, Jeon ES, Kim MS, Hwang KK, Chae SC, Baek SH, Kang SM, Choi DJ, Yoo BS, Kim KH, Cho MC, Kim JJ, Oh BH. Reverse J-Curve Relationship Between On-Treatment Blood Pressure and Mortality in Patients With Heart Failure. JACC Heart Fail. 2017 Nov;5(11):810-819. doi: 10.1016/j.jchf.2017.08.015. PMID 29096790
- [Derived] Lee H, Lee SE, Park CS, Park JJ, Lee GY, Kim MS, Choi JO, Cho HJ, Lee HY, Choi DJ, Jeon ES, Kim JJ, Oh BH. Hyponatraemia and its prognosis in acute heart failure is related to right ventricular dysfunction. Heart. 2018 Oct;104(20):1670-1677. doi: 10.1136/heartjnl-2017-312084. Epub 2017 Oct 27. PMID 29079633